CLINICAL TRIAL: NCT03824886
Title: Enhancing SKIN Health and Safety in Aged CARE: An Exploratory Cluster Randomized Pragmatic Trial in Aged Nursing Home Residents (SKINCARE)
Brief Title: Enhancing SKIN Health and Safety in Aged CARE
Acronym: SKINCARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PD Dr. Jan Kottner (Other)
Responsible Party: Sponsor-Investigator, PD Dr. Jan Kottner, Scientific Director Clinical Research Center for Hair and Skin Science, Charite University, Berlin, Germany
Organization: Charite University, Berlin, Germany (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CRC-SP-A-30
Record Dates: First submitted 2019-01-21; First posted 2019-01-31 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-08

CONDITIONS: Xerosis Cutis; Dry Skin; Pruritus; Pressure Ulcer; Intertrigo; Incontinence-associated Dermatitis; Skin Tear; Skin Care
Keywords: Skin Integrity; Aged Care Receivers; Care Dependent; Geriatric Patients; Prevention; Skin Protection
MeSH Terms: conditions — Pruritus; Pressure Ulcer; Intertrigo

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Implementation of skin care algorithm (Experimental): In the interventional nursing homes, a structured skin care prevention package based on a newly developed evidence-based skin care algorithm will be implemented at the nursing homes and delivered by nurses.
  Interventions: Other: Implementation of skin care algorithm
- Standard Care (No Intervention): In the control group, no additional intervention will be implemented. PU and IAD prevention and basic hygiene and skin care activities are routinely conducted in German nursing homes. This is considered as 'usual practice'.

INTERVENTIONS:
Other: Implementation of skin care algorithm — Implementation of structured and standardized skin care regimen
  Arms: Implementation of skin care algorithm

SUMMARY:
Aged long-term care receivers are affected by various adverse skin conditions like pressure ulcers, incontinence-associated dermatitis, dryness, intertrigo and many more. Prevention of these skin problems and the provision of general hygiene and skin care activities are key areas of nursing practice. Numerous condition specific guidelines are available and are implemented separately. The more guidelines exist, the more difficult it is for nurses to implement them all. On the other hand, there is a huge overlap in terms of aetiology, pathogenesis and prevention of aforementioned skin conditions.

The overall aim of this trial is to test the feasibility and to estimate possible effects of a comprehensive skin care package targeting main nursing relevant skin problems at the same time. Therefore a study will be performed in nursing homes of the state of Berlin comparing the skin care package to standard care. Residents' safety and subjective wellbeing will increase combined with improvements in professional competence of nurses. An advisory board consisting of international experts agreed already to supervise the trial.

DETAILED DESCRIPTION:
Objectives and aims:

Aged and care dependent patients suffer from many adverse skin conditions like xerosis cutis (including pruritus), pressure ulcers, skin tears, intertrigo and incontinence-associated dermatitis. Separate preventive strategies for these particular risks and diseases are available and partly implemented. Although distinct clinical diagnoses, there are substantial overlaps in terms of etiology (e.g. skin fragility, immobility) pathophysiology, prevention (e.g. safe handling, off-loading) and treatment (e.g. skin protection and care). Facilities are challenged to implement fragmented, condition-specific guidelines, neglecting shared etiologies and prevention and treatment principles, which has been shown to be an important barrier for implementation of evidence-based practice.

Recently an evidence-based comprehensive skin care algorithm was developed. The objective of this trial is to investigate the feasibility of the implementation of this skin care package, to describe context factors for implementation, to estimate effect sizes and intracluster coefficients.

Study design:

An exploratory cluster randomized trial in aged nursing home residents will be conducted. The cluster design was chosen to avoid contamination between groups. A total of n = 500 residents from n = 20 nursing homes (randomly selected from the population of nursing homes of the state of Berlin) will be included in the study. In the intervention group (n = 10 nursing homes), the developed evidence-based algorithm will be implemented. The control group (n = 10 nursing homes) receives the usual standard care of the respective nursing home.

ELIGIBILITY:
Inclusion/ Exclusion Criteria for Residents:

Inclusion Criteria:

* Living in the nursing home,
* 65+ years,
* 'Care degree 2' or higher according to SGB XI (Sozialgesetzbuch (Codebook of Social Law)),
* Written informed consent (by legal representative if required)

Exclusion Criteria:

* Residents at end of life,
* Any dermatological condition or skin affection requiring dermatological treatment,
* Known allergies to any product ingredients

Inclusion/ Exclusion Criteria for Nursing Homes:

Inclusion Criteria:

* Nursing home in the federal state of Berlin with at least n = 70 or more residents.
* Expression of a clear commitment to implement the skin care algorithm if assigned to the intervention group,
* Valid pressure ulcer prevention standard/algorithm is in place,
* Written commitment to adherence to the trial procedures regardless of the outcome of randomisation. Exclusion criteria:
* Nursing homes with less than n = 70 residents in the federal state of Berlin.

Exclusion Criteria:

* Nursing homes with less than n = 70 residents in the federal state of Berlin

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 405 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2021-06-04 (Actual); Study Completion 2021-06-04 (Actual)

PRIMARY OUTCOMES:
Incidence of Pressure Ulcers (PU) Category II, III, IV, Unstageable, Deep Tissue Injury (DTI) | Week 12 +/- 1
  Proportions of newly developed PUs per person and per skin area to calculate the cumulative incidence
Incidence of Pressure Ulcers (PU) Category II, III, IV, Unstageable, Deep Tissue Injury (DTI) | Week 24 +/- 1
  Proportions of newly developed PUs per person and per skin area to calculate the cumulative incidence
Location of Pressure Ulcers (PU) Category II, III, IV, Unstageable, Deep Tissue Injury (DTI) | Week 12 +/- 1
  Classification according to NPUAP (National Pressure Ulcer Advisory Panel)/EPUAP (European Pressure Ulcer Advisory Panel) 2014
Location of Pressure Ulcers (PU) Category II, III, IV, Unstageable, Deep Tissue Injury (DTI) | Week 24 +/- 1
  Classification according to NPUAP (National Pressure Ulcer Advisory Panel)/EPUAP (European Pressure Ulcer Advisory Panel) 2014
Incidence of Incontinence-associated Dermatitis (IAD) | Week 12 +/- 1
  Proportions of newly developed IAD per person and per skin area to calculate the cumulative incidence. The classification of IAD will be according to GLOBIAD (Ghent Global IAD Categorisation tool) and distinction between intact and eroded skin according to Proceedings of the Global IAD Expert Panel.
Incidence of Incontinence-associated Dermatitis (IAD) | Week 24 +/- 1
  Proportions of newly developed IAD per person and per skin area to calculate the cumulative incidence. The classification of IAD will be according to GLOBIAD (Ghent Global IAD Categorisation tool) and distinction between intact and eroded skin according to Proceedings of the Global IAD Expert Panel.
Incidence of Intertrigo | Week 12 ± 1
  Proportions of newly developed intertrigo per person and skin area to calculate the cumulative incidence. Medical diagnoses according to ICD (international classification of diseases) 11.
Incidence of Intertrigo | Week 24 ± 1
  Proportions of newly developed intertrigo per person and skin area to calculate the cumulative incidence. Medical diagnoses according to ICD (international code of diseases) 11.
Incidence of Skin Tears (ST) | Week 12 ± 1
  Proportions of newly developed STs per person and skin area to calculate the cumulative incidence. Classification according to ISTAP (International Skin Tear Advisory Panel).
Incidence of Skin Tears (ST) | Week 24 ± 1
  Proportions of newly developed STs per person and skin area to calculate the cumulative incidence. Classification according to ISTAP (International Skin Tear Advisory Panel).

SECONDARY OUTCOMES:
Overall Dry Skin Score (ODS) on face, trunk, arms, hands, feet, legs | Week 0, Week 12 ± 1, Week 24 ± 1
  Change in Overall Dry Skin score. ODS is a clinical assessment of the presence and severity of skin dryness using a five-point scale. A score of '0' indicates no skin dryness, whereas a score of '4' indicates advanced skin roughness, large scales, inflammation and cracks.
Stratum Corneum Hydration (SCH) measurements on right lower leg lateral, right midvolar forearm | Week 0, Week 12 ± 1, Week 24 ± 1
  Change in Stratum Corneum Hydration. SCH was measured using the Corneometer CM 825 (Courage + Khazaka, Cologne, Germany). This measurement is based on the differences of the dielectric constant of water and other substances. With this device, only the moisture content in the stratum corneum is measured. The arbitrary units (a.u.) range from 0 to 120 where as higher readings indicate higher stratum corneum hydration.
  * Means of triplicate measurements per skin area in arbitrary units at right lower leg lateral, right midvolar forearm
  * If measurements are not possible at right leg/arm (e.g. due to amputation) they will be conducted at contralateral skin areas
Transepidermal Water Loss (TEWL) on right lower leg lateral, right midvolar forearm | Week 0, Week 12 ± 1, Week 24 ± 1
  Change in Transepidermal water loss. TEWL was measured with the Tewameter TM 300 (Courage + Khazaka, Cologne, Germany). The probe captures the constant permeation of water through the stratum corneum in gram per hour per m2. The measuring probe contains a pair of sensors that are located in different distances to the skin surface to determine temperature and relative humidity above the skin surface. The humidity gradient between both sensors is used for calculating the transepidermal water loss. Higher values indicate a higher transepidermal water loss.
  * Means of duplicate measurements per skin area in g/m2/h at right lower leg lateral, right midvolar forearm
  * If measurements are not possible at right leg/arm (e.g. due to amputation) they will be conducted at contralateral skin areas
Skin Surface pH on right lower leg lateral, right midvolar forearm | Week 0, Week 12 ± 1, Week 24 ± 1
  Change in Skin surface pH. Skin surface pH was measured with the Skin-pH-Meter PH 905 (Courage + Khazaka, Cologne, Germany), a planar glass electrode. The pH is a measure of acidity and alkalinity of a solution and it indicates the concentration of the hydrogen ions in an aqueous solution. Reference values of human skin have been reported to range from 4 to 6.
  * Means of duplicate measurements per skin area at right lower leg lateral, right midvolar forearm
  * If measurements are not possible at right leg/arm (e.g. due to amputation) they will be conducted at contralateral skin areas
Skin surface temperature [°C] on right lower leg lateral, right midvolar forearm | Week 0, Week 12 ± 1, Week 24 ± 1
  Skin surface temperature was measured with the Skin-Thermometer ST 500 (Courage+Khazaka electronic GmbH).
  * Means of duplicate measurements per skin area in °C at right lower leg lateral, right midvolar forearm
  * If measurements are not possible at right leg/arm (e.g. due to amputation) they will be conducted at contralateral skin areas
Quality of Life (QoL) (residents without cognitive impairment): WHO-Five Well-being Index (WHO = World Health Organization) | Week 0, Week 24 ± 1
  Self-completion of the WHO-Five Well-being Index by residents without cognitive impairment. The German version of the WHO-Five Well-being Index questionnaire published by the World Health Organization in 1998 will be used. Scores range from '5' (all the time) to '0' (never) for in total five items.The sum scores range from 0, indicating the lowest well-being, to 25, indicating the highest well-being. A cut-off score of < 13 is recommended. Means will be calculated.
  ◦ Means
Quality of Life (QoL) (cognitively impaired residents): QUALIDEM 18-Item Assessment (QUALIDEM = No original term, measurement instrument for proxy rating of quality of life in people with dementia) | Week 0, Week 24 ± 1
  The QUALIDEM assessment is a dementia-specific quality of life (QoL) instrument carried out by the nursing staff that allows a proxy-based QoL rating in all stages of dementia.The German version of the QUALIDEM version 2.0 published in 2015 will be used.Residents with a very severe dementia will answer the 18-item Instrument.To assess whether the resident is affected by mild to severe dementia or very severe dementia the global deterioration scale (GDS) will be used (see Outcome 22).
Quality of Life (QoL) (cognitively impaired residents): QUALIDEM 37-Item Assessment | Week 0, Week 24 ± 1
  The QUALIDEM assessment is a dementia-specific quality of life (QoL) instrument carried out by the nursing staff that allows a proxy-based QoL rating in all stages of dementia.The German version of the QUALIDEM version 2.0 published in 2015 will be used.In case the resident is affected by a mild to severe dementia the 37-item assessment will be used.To assess whether the resident is affected by mild to severe dementia or very severe dementia the global deterioration scale (GDS) will be used (see Outcome 22).
Itch Assessment | Week 0, Week 12 ± 1, Week 24 ± 1
  * Self-completion of the 5-D itch scale by residents without cognitive impairment (according to GDS score of 1)
  * The score of the 5-D Itch scale ranges from '5' (no pruritus) to '25' (most severe pruritus) and contains five items measuring pruritus over the past two weeks.
  * Means
Pain Assessment (residents without cognitive impairment): numeric rating scale | Week 0, Week 12 ± 1, Week 24 ± 1
  ◦ Self-completion of a numeric rating scale (NRS with total scores from 0: minimum pain to 10: maximum pain) to measure pain by residents without cognitive impairment. Means of the total score will be calculated.
Pain Assessment (cognitively impaired residents): Verbal rating scale | Week 0, Week 12 ± 1, Week 24 ± 1
  ◦ Verbal rating scale (proxy rated) to measure pain in cognitively impaired residents (VRS with total scores from 0: minimum pain to 10: maximum pain). Means of the total score will be calculated.
Assesment of dementia: Global Deterioration scale. | Week 0
  To assess whether the resident is affected by mild to severe dementia or very severe dementia the global deterioration scale (GDS) will be used. GDS scores from 2 to 6 indicate a mild to severe dementia and the 37-item assessment of the QUALIDEM tool will be used (see Outcome 18). A GDS score of 7 indicates very severe dementia and the 18-item QUALIDEM tool will be used (see Outcome 17).

CONTACTS AND LOCATIONS:
Overall Officials: Jan Kottner, Prof. Dr., Principal Investigator — Charite University, Berlin, Germany
Locations (2):
- Germany (2):
  - Charité - Universitätsmedizin Berlin, Berlin
  - Charité-Universitätsmedizin Berlin, Berlin

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Amin R, Volzer B, El Genedy-Kalyoncu M, Blume-Peytavi U, Kottner J. Skin care types, frequencies and products: A cross-sectional study in German institutional long-term care. J Tissue Viability. 2024 May;33(2):318-323. doi: 10.1016/j.jtv.2024.02.005. Epub 2024 Feb 10. PMID 38360494
- [Derived] Volzer B, El Genedy-Kalyoncu M, Fastner A, Tomova-Simitchieva T, Neumann K, Hillmann K, Blume-Peytavi U, Hahnel E, Sill J, Balzer K, Kottner J. Enhancing skin health and safety in aged care (SKINCARE trial): A cluster-randomised pragmatic trial. Int J Nurs Stud. 2024 Jan;149:104627. doi: 10.1016/j.ijnurstu.2023.104627. Epub 2023 Oct 28. PMID 37956524
- [Derived] Volzer B, El Genedy-Kalyoncu M, Fastner A, Tomova-Simitchieva T, Neumann K, Sill J, Balzer K, Kottner J. Prevalence and associations of xerosis cutis, incontinence-associated dermatitis, skin tears, pressure ulcers, and intertrigo in aged nursing home residents: A representative prevalence study. Int J Nurs Stud. 2023 May;141:104472. doi: 10.1016/j.ijnurstu.2023.104472. Epub 2023 Feb 23. PMID 36898269
- [Derived] Kottner J, Hahnel E, El Genedy M, Neumann K, Balzer K. Enhancing SKIN health and safety in aged CARE (SKINCARE Trial): a study protocol for an exploratory cluster-randomized pragmatic trial. Trials. 2019 May 29;20(1):302. doi: 10.1186/s13063-019-3375-7. PMID 31142364